CLINICAL TRIAL: NCT03629847
Title: Treatment of Neuroendocrine Tumors (NETs) With Combination of Everolimus and Radiolabeled Somatostatin Analogue
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2121-159
Record Dates: First submitted 2013-09-30; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Neuroendocrine Tumors
Keywords: NETs, MTD, Everolimus.
MeSH Terms: conditions — Neuroendocrine Tumors; Metatropic dwarfism | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus & Radiolabeled Lu-177 (Experimental): Drug: Everolimus will be administrated in combination with the intravenous radiolabelled Lu-177 DOTATATE therapy.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Drug: Everolimus will be administrated in combination with the intravenous radiolabelled Lu-177 DOTATATE therapy.
  Other Names: Radiolabeled Lu-177 DOTATATE

SUMMARY:
NET originate in neuroendocrine cells throughout the body. The goal of this study is to assess the safety and efficacy of the combination of everolimus and the intravenous radiolabeled Lu-177 DOTATATE Therapy as a 1st line therapy in unresectable well to moderately differentiated metastatic neuroendocrine tumors of all GI, lung and pancreatic origins. This is a phase 1 - 2 study. The phase 1 part involves finding the maximum tolerating dose (MTD) of Everolimus.

DETAILED DESCRIPTION:
Neuroendocrine tumors NET refers to tumors that originate in neuroendocrine cells throughout the body (including in the thymus, lung, pancreas, gastrointestinal [GI] tract and less common sites). They can be broadly subclassified into well-differentiated and poorly differentiated cancers. Treatment of well differentiated NET are complex and involves surgical, Locoregional and systemic modalities depending on the manifestations as well as extent of disease. Treatment is best planned in a multidisciplinary tumor board. Of the emerging new systemic modalities are Everolimus and radiolabelled somatostatin analogue. The goal of this study is to assess the safety and efficacy of the combination of everolimus and the intravenous radiolabeled Lu-177 DOTATATE Therapy (a somatostatin analogue) as a first line therapy in unresectable well to moderately differentiated metastatic neuroendocrine tumors of all gastrointestinal, lung and pancreatic origins. This is a phase 1 - 2 study. The phase 1 part involves finding the maximum tolerating dose (MTD) of Everolimus.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Histologically confirmed well to moderately differentiated neuroendocrine tumors of GI, lung or pancreatic origin. The grading follows the WHO grading system (Appendix III).
* Measurable disease by CT or MRI.
* Positive Tc-99m Octreotide scan or Ga-68 Octreotate scan (Positive means uptake at tumor sites).
* Advanced disease which are not treatable by surgical resection.
* Documented progressive disease within the past 12 months.
* WHO Performance Status 0 - 2.
* Fasting blood sugar ≤ 1.5 Χ Upper Limit of Normal (ULN).
* Fasting triglycerides ≤ 2.5 Χ Upper Limit of Normal (ULN), and fasting cholesterol ≤ 300 mg/dl or ≤ 7.75 ml/l.
* Adequate renal function with creatinine clearance ≥ 60 ml/l.
* Adequate hepatic function:
* Total bilirubin ≤ 1.5 Χ Upper Limit of Normal (ULN)
* Liver Function Tests (Serum aspartate aminotransferase and alanine transaminase levels) ≤ 2.5 Χ ULN (and ≤ 5 Χ ULN, in case of presence of liver metastasis)
* Adequate hematological values:
* Absolute neutrophil count ≥ 1 x 109/L
* Platelet count ≥ 100 x 109/L
* Signed written informed consent before enrolment.

Exclusion Criteria:

* Readily completely Resectable disease.
* Prior therapy with everolimus or systemic chemotherapy.
* Prior chemoembolization, radio-embolization, or bland embolization within 6 months before enrolment. Likewise, patients are ineligible if had undergone conventional radiotherapy, radiofrequency ablation, cryoablation or alcohol injection within 1 month prior to enrolment.
* Prior long acting somatostatin analogue within 1 month prior to enrolment. Short acting somatostatin analogue is allowed as long as it is not administered within 12 hours before or /and 12 hours after the administration of the intravenous radiolabelled Lu-177 DOTATATE Therapy.
* Presence of Central Nervous System metastasis.
* Previous malignancy within 5 years, except adequately treated non melanomatous skin cancer or in situ cervical cancer
* Other active malignancy.
* HIV infection.
* Severe or uncontrolled medical conditions, such as:
* Active uncontrolled severe infection
* History of invasive fungal infection.
* Child C liver dysfunction.
* Severely impaired lung function.
* Psychiatric or mental disorder, precluding understanding of the information of the trial related topics and giving valid informed consent.
* Any psychological, familial, geographic or social circumstances which could impair the patient's ability to participate in the trial and comply with follow up.
* Treatment with other anti-cancer therapy.
* Known hypersensitivity to any of the study drugs.
* Pregnant or breast feeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | "3 years"
  Establish safety profile of the combination of everolimus and intravenous radiolabeled Lu-177 DOTATATE

SECONDARY OUTCOMES:
Survival assessment | 3 years
  Progression free survival (PFS) and Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Aljubran, MD, Principal Investigator — KFSH&RC; Fazal Hussain, MD, Study Director — KFSH&RC
Locations (1):
- Oncology Centre, King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided